CLINICAL TRIAL: NCT03278002
Title: Uptravi® (SelexiPag): tHe usErs dRug rEgistry
Brief Title: A Registry for Patients Taking Uptravi
Acronym: SPHERE
Status: Completed | Type: Observational
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Other Study IDs: AC-065A402
Record Dates: First submitted 2017-08-29; First posted 2017-09-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group/Cohort Information: This is a US multi-center, prospective, real world, observational drug registry enrolling patients actively treated with Uptravi. Participating patients will be followed prospectively for a maximum of 18 months from the date of enrollment into the registry.

SUMMARY:
This is a US multi-center, prospective, real world, observational drug registry enrolling patients actively treated with Uptravi. Participating patients will be followed prospectively for a maximum of 18 months from the date of enrollment into the registry.

ELIGIBILITY:
Inclusion Criteria:

* Signed patient informed consent form (ICF).
* Patients ≥ 18 years of age at time of Uptravi initiation, and
* Patients who initiate Uptravi:

  * at enrollment, or
  * less than or equal to 60 days prior to enrollment and have a documented titration regimen (defined as all documented dose changes including, but not limited to: starting dose and dates and highest tolerated dose and dates)

Exclusion Criteria:

* Patients previously exposed to Uptravi treatment during a clinical trial.
* Patients that previously discontinued Uptravi for any reason, prior to study enrollment (discontinuation defined as an interruption of therapy greater than or equal to 30 days).
* Patients enrolled in a blinded clinical trial or in a clinical trial involving an unapproved drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The number of patients planned to be enrolled in the study is approximately 800 patients from approximately 80 centers in the U.S.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Using Electronic Medical Records, the change in Hemodynamics (by Right Heart Catherization), WHO FC and 6 Minute Walk Distance (by meters) from diagnosis to registry enrollment and to EOS will be measured/collected. | Followed prospectively for a maximum of 18 months from the date of enrollment into the registry.
  To describe demographics and disease characteristics of patients treated with Uptravi.
The initial dose (in micrograms), dose at selected intervals (in days), highest dose, maintenance dose, time between titrations, time from initiation to maintenance dose (in days) and total duration of exposure to Uptravi (in days) will be collected. | Followed prospectively for a maximum of 18 months from the date of enrollment into the registry.
  To describe the dosing regimens and titration of Uptravi, including any transition from other PAH specific therapies to Uptravi and from Uptravi to other prostanoids.
Occurrence of AEs and SAEs (incl. hospitalizations), discontinuation of Uptravi and reason for stopping and occurrence of all-cause death by relationship to PAH. | Followed prospectively for a maximum of 18 months from the date of enrollment into the registry.
  To describe the clinical course of patients treated with Uptravi.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion, Study Director — Actelion
Locations (85):
- United States (84):
  - University of South Alabama, Mobile, Alabama
  - Pulmonary Associates, Phoenix, Arizona
  - Cardioivascular Consultants, Ltd., Phoenix, Arizona
  - University of Arizona-Clinical Translational and Regenerative Medicine, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - VA Greater Los Angeles Healthcare Center, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA, Torrance, California
  - University of Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - Banner Health Research Institute, Greeley, Colorado
  - Florida Lung Asthma and Sleep Specialists, Celebration, Florida
  - Broward Pulmonary and Sleep, Fort Lauderdale, Florida
  - University of Florida, HSC, Gainesville, Florida
  - West Pasco Pulmonary Associates, Hudson, Florida
  - University of Florida-Jacksonville College of Medicine, Jacksonville, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Wellstar Marietta Pulmonary Medicine, Marietta, Georgia
  - University of Chicago Hospitals, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - CIC Associates, Clive, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Oschner Clinic Foundation/Oschner Medical Center, New Orleans, Louisiana
  - Chest Medicine Associates, South Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Tufts University Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Research, Mercy Hospital Saint Louis, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Pulmonary Health Physicians, PC, Fayetteville, New York
  - Winthrop University Hospital, Mineola, New York
  - Northwell Health, New Hyde Park, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weil Cornell Medicine, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina Hospitals at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - Legacy Medical Group-Pulmonary and Sleep Clinic, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health Medical Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott and White Health, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas, Houston Health Center, Houston, Texas
  - Methodist Healthcare of San Antonio, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax, Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Providence Health & Services d/b/a/ Providence Sacred Heart Medical Center & Children's Hospital Providence Medical Research Center, Spokane, Washington
  - Multicare Institute for Research & Innovation, Tacoma, Washington
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin
  - Aurora Research Institute / Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- CardioPulmonary Research, PSC, Guaynabo, Puerto Rico

REFERENCES:
- [Derived] Kim NH, Hemnes AR, Chakinala MM, Highland KB, Chin KM, McLaughlin V, Zhao C, Narayan V, Farber HW. Patient and disease characteristics of the first 500 patients with pulmonary arterial hypertension treated with selexipag in real-world settings from SPHERE. J Heart Lung Transplant. 2021 Apr;40(4):279-288. doi: 10.1016/j.healun.2021.01.006. Epub 2021 Jan 15. PMID 33526303